CLINICAL TRIAL: NCT05047614
Title: Effects of Lumbar Repositioning Feedback and Transversus Abdominis Training on Lumbar Propricption in Patients With Chronic Mechanical Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mai Hassan Ahmed Desouki, Assistant Lecturer, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 153145
Record Dates: First submitted 2020-07-22; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study 1 (Experimental): Twelve patients in study group 1 receiving lumbar repositioning feedback training
  Interventions: Device: including sham
- Study 2 (Experimental): Twelve patients in study group 2 receiving transverses abdominis training
  Interventions: Device: including sham
- Study 3 (Experimental): Twelve patients in study group 3 receiving both lumbar repositioning feedback training and tranversus abdominis training
  Interventions: Device: including sham
- Control (Experimental): Twelve patients in control group receiving conventional lumbar propriception physical therapy program .
  Interventions: Device: including sham

INTERVENTIONS:
Device: including sham — Repositiong feedback training and biofeedback pressure training unit

SUMMARY:
This study is conducted to answer the following question: What is the effect of lumbar repositioning feedback and transverses abdominis training on lumbar proprioception in patients with chronic mechanical low back pain?

DETAILED DESCRIPTION:
Chronic low back pain is a chronic pain syndrome in the lower back region, lasting for at least twelve weeks. Chronic low back pain represents the leading cause of disability worldwide and is a major welfare and economic problem. Low back pain represents a major social and economic problem. The prevalence of chronic low back pain is estimated to range from fifteen to forty-five percent in French healthcare workers. Low back pain symptoms can derive from many potential anatomic sources, such as nerve roots, muscle, fascial structures, bones, joints, intervertebral discs, and organs within the abdominal cavity. Moreover, symptoms can also spawn from aberrant neurological pain processing causing neuropathic low back pain. Low back pain has been associated with motor control dysfunction. Indicators of this dysfunction include decreased contraction of the transversus abdominis and multifidus muscles, the reduced cross-sectional area of the multifidus, and fat infiltration. An association of chronic low back pain with altered muscle recruitment patterns and transversus abdominis activation delay was also found, as well as increased back muscle fatigue and altered kinematic patterns in the hips and lumbar area.

This was further supported in two recent systematic reviews that reported that proprioception deficits were found in patients with chronic low back pain compared to healthy controls

ELIGIBILITY:
Inclusion Criteria:

* Patients with CMLBP referred from orthopedic surgeon with no radicular pain
* Their age is ranged between 35-55 years old (Martim etal.,2008)
* BMI 24-28 kg/m2

Exclusion Criteria:

* Patients who have a history of diabetic peripheral neuropathies
* Patients who have a history of sciatica
* Spinal or lower limb deformity or any pathology within the spine.
* Patients who have neurological disorders
* Patients who have a history of previous lumbar surgery
* Patients who have visual problems

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-04-19 (Actual); Primary Completion 2022-05-02 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Pressure biofeedback unit | up to 45 days
  Assessment of transversus abdominis activation
feedback laser tracker | up to 45 days
  Assessment of lumbar repositioning error

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No